CLINICAL TRIAL: NCT02793141
Title: International, Multi Centre, Prospective, Observational Cohort Study of Nosocomial Pneumonia in Intensive Care Units
Brief Title: International Study on NoSocomial Pneumonia in Intensive CaRE (PneumoINSPIRE)
Acronym: PneumoINSPIRE
Status: Completed | Type: Observational
Sponsor: The University of Queensland (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Despoina Koulenti, MD, PhD, Research Fellow, The University of Queensland
Other Study IDs: 2015000302
Record Dates: First submitted 2016-05-22; First posted 2016-06-08 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Nosocomial Pneumonia
Keywords: Pneumonia; Intensive Care Unit; Nosocomial pneumonia; Hospital-acquired pneumonia; Ventilator-associated pneumonia; ICU; HAP; VAP; Critical Care
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICU Nosocomial Pneumonia: Nosocomial pneumonia (hospital-acquired pneumonia) with onset in non-intubated ward patients (= or > 48 hours after hospital admission) that due to deterioration are subsequently admitted to ICU or nosocomial pneumonia (hospital-acquired pneumonia) with onset in non-intubated ICU patients (= or >48 hours after hospital admission) or ventilator-associated pneumonia with onset = or > 48 hours after intubation. No intervention will be administered.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be administered

SUMMARY:
The International study on NoSocomial Pneumonia in Intensive CaRE (PneumoINSPIRE) is a prospective, international, multicentre, observational, cohort study. The study aims to provide up-to-date and generalisable information on current worldwide epidemiology and clinical practice associated with diagnosis and management of nosocomial pneumonia in Intensive Care Unit (ICU) patients.

PneumoINSPIRE study is endorsed by the European Society of Intensive Care Medicine (ESICM).

DETAILED DESCRIPTION:
Specifically, the study aims to:

* Evaluate the global epidemiology of nosocomial pneumonia in ICU patients, analysing responsible pathogens and resistance pattern by type of pneumonia and geographical region.
* Describe on a global scale current clinical practice regarding diagnosis and determine the degree of concordance between the diagnosis of nosocomial pneumonia in routine clinical practice and the official definitions including: a) ATS/IDSA 2005 guidelines; b) CDC/NHSN Surveillance Definitions (version January 2015, modified April 2015).
* Identify on a global scale variable treatment decisions with emphasis on therapeutic schemas, appropriateness, de-escalation decisions and their relation to outcomes.

Secondary objectives include:

* Evaluate nosocomial pneumonia in specific subgroups of critically ill patients (such as, chronic obstructive pulmonary disease [COPD], the elderly, postoperative, trauma patients).
* Describe the differences between nosocomial pneumonia in non-intubated ICU patients and VAP.
* Compare the characteristics and outcomes between patients with nosocomial pneumonia in ward patients later transferred to the ICU and non-intubated ICU patients with nosocomial pneumonia.

This international study will explore clinical details for nosocomial pneumonia in the ICU setting: practice variations among countries and continents, diagnostic and treatment modalities, implicated pathogens and their resistance patterns, resolution patterns and risk factors for unfavourable outcomes. In view of these, this global multicentre study shall provide useful information for the elaboration of future recommendations on diagnostic and treatment approaches for nosocomial pneumonia in the ICU.

Inclusion criteria:

ICU patients with a diagnosis of nosocomial pneumonia, including:

* Admission to the ICU with diagnosis of HAP that developed in the ward in non-intubated patients (Ward HAP)
* The first episode of ICU-acquired pneumonia that developed in non-intubated patients (ICU-HAP)
* The first episode of ICU-acquired pneumonia that developed in patients receiving invasive ventilation(i.e. Ventilator-Associated Pneumonia (VAP)).

Exclusion criteria:

* Age < 18 years
* Patients with nosocomial pneumonia receiving palliative treatment at the time of assessment for eligibility (i.e. the time of clinical diagnosis)
* Previous inclusion in the study

Research sites:

More than 150 ICUs from 25 or more countries worldwide that will agree to participate in the study.

Sample size:

A minimum of 10 consecutive ICU patients with nosocomial pneumonia as described above will be recruited per site. A sample size of at least 1000 ICU patients with nosocomial pneumonia is anticipated to comprise the dataset. This sample size has been chosen to provide generalisable data for each geographic region and to satisfy power considerations.

Statistical analysis:

Descriptive analytic, techniques and parametric and non-parametric tests will be used to explore diagnostic, microbiological or subgroup differences as well as clinical outcomes of nosocomial pneumonia. Cox regression will be used to predict dichotomous outcomes of interest, including mortality and pneumonia resolution. Independent predictors and associated hazard ratios with 95% confidence intervals will be reported. A two-sided p-value less than 0.05 will be considered statistically significant.

Proposed Start and End Date:

The first site is anticipated to commence recruitment in March 2016 with staggered site recruitment; however, sites are anticipated to start recruitment during the first half of 2016; each site will commence recruitment as soon as relevant Institutional Review Board approvals have been obtained. Recruitment will continue until the minimum target of 10 patients has been reached. Sites will have the opportunity for further recruitment while the study is active. Completion of recruitment is anticipated to occur by end December 2018.

Dissemination of Findings:

Summary data will be presented in a timely manner at national and international conferences and in peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

ICU patients with a diagnosis of nosocomial pneumonia, including:

* Admission to the ICU with diagnosis of HAP that developed in the ward in non-intubated patients (Ward HAP)
* The first episode of ICU-acquired pneumonia that developed in non-intubated patients
* The first episode of ICU-acquired pneumonia that developed in patients receiving invasive ventilation (i.e. Ventilator-Associated Pneumonia (VAP)).

Exclusion Criteria:

* Age < 18 years
* Patients with nosocomial pneumonia receiving palliative treatment at the time of assessment for eligibility
* Previous inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every ICU that will agree to participate to the study and receive ethics approval (or waiver of need for ethics approval) according to the local and national regulations in each country.
  Every ICU patient with the diagnosis of nosocomial pneumonia hospitalised in the ICU.
  Every patient with the above diagnosis, > or = 18 years old, not receiving palliative treatment at the time of assessment for eligibility, not previously included in the study and fulfilling the inclusion criteria is eligible.
Sampling Method: Non-Probability Sample
Enrollment: 1657 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Mortality | Day 28
  ICU and hospital mortality, censored at Day 28 if ICU discharge is later than day 28. Day 1 is the day of onset for pneumonia with arises in the ICU and day of ICU admission for pneumonia without ICU onset.
Degree of concordance of clinical diagnosis of VAP with official definitions | Day 28 or ICU discharge, whichever occurs first
  The degree of concordance with diagnosing nosocomial pneumonia with:
  1. ATS/IDSA 2005 Guidelines
  2. CDC/NHSN Surveillance definitions (Jan 2015, modified April 2015)
Pathogenic organism (categorical) | Day 28 or ICU discharge, whichever occurs first
  Responsible pathogens and resistance pattern by type of pneumonia and geographical region (% per category)
Clinical management of pneumonia (categorical) | Day 28 or ICU discharge, whichever occurs first
  Empirical management, modification of empirical management (escalation, de-escalation and discontinuation) and duration of antibiotic treatment for pneumonia
Resolution of pneumonia (categorical) | Day 3, 7 and 14
  Clinical resolution of the pneumonia at pre-selected time periods

SECONDARY OUTCOMES:
Recurrence of pneumonia | Day 14 and 28
  Clinical recurrence of the pneumonia within a set period of time
Mechanical ventilation-free days | Censored at Day 28 or discharge from ICU, whichever occurs first
  Number of days the patient does not require mechanical ventilation whilst in ICU and censored at Day 28
Number of antibiotic-free days | Censored at Day 28 or discharge from ICU, whichever occurs first
  Number of days patient did not require antibiotic therapy whilst in ICU and censored at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Despoina Koulenti, MD,PhD, Principal Investigator — Post-doctoral Research Fellow, Burns Trauma and Critical Care Research Centre, Faculty of Medicine, The University of Queensland; Jeffrey Lipman, MBBCh, MD, Study Director — Director of Burns Trauma and Critical Care Research Centre, School of Medicine, The University of Queensland
Locations (2):
- Royal Brisbane and Womens Hospital (RBWH), Brisbane, Australia
- University Critical Care Department, Aghioi Anargyroi Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koulenti D, Armaganidis A, Arvaniti K, Blot S, Brun-Buisson C, Deja M, De Waele J, Du B, Dulhunty JM, Garcia-Diaz J, Judd M, Paterson DL, Putensen C, Reina R, Rello J, Restrepo MI, Roberts JA, Sjovall F, Timsit JF, Tsiodras S, Zahar JR, Zhang Y, Lipman J; Working Group on Pneumonia of the European Society of Intensive Care Medicine. Protocol for an international, multicentre, prospective, observational study of nosocomial pneumonia in intensive care units: the PneumoINSPIRE study. Crit Care Resusc. 2023 Oct 18;23(1):59-66. doi: 10.51893/2021.1.OA5. eCollection 2021 Mar. PMID 38046390